CLINICAL TRIAL: NCT07404462
Title: Correlation Between Tumor-infiltrating Lymphocytes and Response to Systemic Therapy in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ERIDKE-0054/2023
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Early Breast Cancer
Keywords: Neoadjuvant Chemotherapy; Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: Single-group study evaluating immune-related tumor stroma factors and circulating biomarkers in patients receiving standard neoadjuvant chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Treatment Group (Experimental): Patients receive standard neoadjuvant chemotherapy according to institutional and international guidelines.
  Interventions: Drug: Neoadjuvant Chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy — Standard neoadjuvant chemotherapy administered according to clinical guidelines.
  Associated Arm(s):

SUMMARY:
This study aims to investigate the correlation between immune-related factors in the tumor stroma and pathological complete response (pCR) in patients with early breast cancer treated with neoadjuvant chemotherapy. In addition, the study evaluates the association between immune-related tumor stroma factors and the presence of circulating tumor cells (CTCs) and circulating tumor DNA (ctDNA) in peripheral blood. The study includes serial blood sampling before and after treatment and during follow-up to assess the prognostic value of these biomarkers for disease progression and recurrence.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy is widely used in patients with early breast cancer to reduce tumor size and improve surgical outcomes. Achieving a pathological complete response (pCR) is associated with improved prognosis; however, reliable predictive biomarkers are still limited. Recent evidence suggests that immune cells in the tumor microenvironment may influence treatment response.

This study evaluates immune-related tumor stroma factors (including tumor-infiltrating lymphocytes and immune marker profiles) in tumor tissue obtained prior to treatment. In parallel, circulating tumor cells (CTCs) and circulating tumor DNA (ctDNA) are assessed from peripheral blood samples collected before neoadjuvant chemotherapy, after completion of treatment, and during follow-up.

The primary objective is to determine whether immune-related tumor stroma factors correlate with pCR after neoadjuvant chemotherapy. Secondary objectives include evaluating the association of immune-related factors with the presence of CTCs and ctDNA and assessing their prognostic value for disease progression and recurrence.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 18 years or older.

Histologically confirmed early breast cancer.

Candidates for standard neoadjuvant chemotherapy.

Ability to provide informed consent.

Exclusion Criteria:

Luminal A subtype of breast cancer.

Prior systemic therapy for breast cancer.

Serious comorbid conditions that would preclude study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | At surgery following completion of neoadjuvant chemotherapy
  Pathological complete response is defined as the absence of invasive carcinoma in the breast and axillary lymph nodes after neoadjuvant chemotherapy (ypT0/Tis ypN0).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No